CLINICAL TRIAL: NCT06750185
Title: A Phase I, First-in-human, Open-label, Dose Escalation Study of the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of BNT317 in Patients With Advanced Solid Tumors
Brief Title: Safety and Preliminary Effectiveness of BNT317, an Investigational Therapy for Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT317-01
Record Dates: First submitted 2024-12-12; First posted 2024-12-27 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumor
Keywords: Malignant solid tumors; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- BNT317 DL1 (Experimental): BNT317 monotherapy
  Interventions: Biological: BNT317 DL1
- BNT317 DL2 (Experimental): BNT317 monotherapy
  Interventions: Biological: BNT317 DL2
- BNT317 DL3 (Experimental): BNT317 monotherapy
  Interventions: Biological: BNT317 DL3
- BNT317 DL4 (Experimental): BNT317 monotherapy
  Interventions: Biological: BNT317 DL4
- BNT317 DL5 (optional, intermediate) (Experimental): BNT317 monotherapy
  Interventions: Biological: BNT317 DL5 (intermediate)
- BNT317 DL6 (optional, intermediate) (Experimental): BNT317 monotherapy
  Interventions: Biological: BNT317 DL6 (intermediate)
- BNT317 DL7 (optional, additional) (Experimental): BNT317 monotherapy
  Interventions: Biological: BNT317 DL7 (additional)

INTERVENTIONS:
Biological: BNT317 DL1 — Intravenous infusion
  Arms: BNT317 DL1
Biological: BNT317 DL2 — Intravenous infusion
  Arms: BNT317 DL2
Biological: BNT317 DL3 — Intravenous infusion
  Arms: BNT317 DL3
Biological: BNT317 DL4 — Intravenous infusion
  Arms: BNT317 DL4
Biological: BNT317 DL5 (intermediate) — Intravenous infusion
  Arms: BNT317 DL5 (optional, intermediate)
Biological: BNT317 DL6 (intermediate) — Intravenous infusion
  Arms: BNT317 DL6 (optional, intermediate)
Biological: BNT317 DL7 (additional) — Intravenous infusion
  Arms: BNT317 DL7 (optional, additional)

SUMMARY:
This is a first-in-human (FIH), open-label, multiple-site, dose escalation study which will evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of increasing doses of BNT317 in participants with advanced solid tumors.

DETAILED DESCRIPTION:
Participants will be assigned to one of four dose levels of BNT317. One treatment cycle contains one treatment.

Participants may receive investigational medicinal product (IMP) for up to 2 years or until they experience disease progression, unacceptable toxicities, withdrawal of consent, study discontinuation or investigator decision. The total duration of the study for a singe participant may be up to 2 years, plus follow-up until the last participant has completed 1 year of survival follow-up (excluding screening).

In the dose escalation phase, an accelerated titration design for Dose Level 1 (DL1) and a Bayesian Optimal Interval (BOIN) design for DL2 to DL4 will be used to evaluate dose limiting toxicities (DLTs) and determine the maximum tolerated dose (MTD).

Additional dosing schedules and/or intermediate or higher dose levels may be evaluated based on the available safety, antitumor activity, PK, and pharmacodynamic (PD) data.

ELIGIBILITY:
Key Inclusion Criteria:

* Have histologically or cytologically confirmed advanced tumors, who have failed standard therapy, or for whom no standard treatment option is available, or for whom standard therapy is not appropriate.
* Have at least one measurable lesion based on RECIST 1.1. Lesions treated after prior local treatment (radiotherapy, ablation, interventional procedures, etc.) are generally not considered as target lesions. If the lesion with prior local treatment is the only targeted lesion, evidence-based radiology must be provided to demonstrate disease progression (the single bone metastasis or the single central nervous system [CNS] metastasis should not be considered as a measurable lesion).
* Adequate hematologic and organ function.

Key Exclusion Criteria:

* Have received any of the following therapies or drugs within the noted time intervals prior to study treatment:

  * Any prior treatment which inhibits cluster of differentiation 39 (CD39).
  * Vaccination with live attenuated vaccine(s) within 4 weeks prior to the first dose of IMP.
  * Any investigational product within 4 weeks or 5 half lives (if the half life of the other investigational product is known), whichever is longer, before the first dose of IMP in this study or ongoing participation in the active treatment phase of another interventional clinical study.
  * Systemic cytotoxic chemotherapy, immunotherapy within 3 weeks or five half-lives of the chemotherapy (whichever is shorter) prior to the first dose of IMP.
  * Radiation therapy (chest, brain or internal organs) within 4 weeks prior to the first dose of IMP.
  * Palliative radiotherapy to metastasis within 2 weeks prior to the first dose of IMP.
  * Systemic corticosteroids (at a dosage greater than 10 mg/day of prednisone or an equivalent dose of other corticosteroids) within 2 weeks prior to the first dose of IMP. Note: local, intranasal, intraocular, intra-articular or inhaled corticosteroids, short term use (≤7 days) of corticosteroids for prophylaxis (e.g., prevention of contrast agent allergy) or treatment of non-autoimmune conditions (e.g., delayed hypersensitivity reactions caused by exposure to allergens) is allowed.
* Have any of the following CNS metastases:

  * Untreated brain metastases that are symptomatic or large (e.g., greater than 2 cm).
  * Treated CNS metastases who are not neurologically stable or on steroids or anticonvulsants within 2 weeks before initiating IMP of this study.
  * Brain metastases treated with radiotherapy that are not confirmed stable by magnetic resonance imaging or contrast-enhanced computer tomography 4 weeks after radiotherapy.
  * Participants with known leptomeningeal metastases.
* Have uncontrolled hypertension or poorly controlled diabetes as specified in the protocol.
* Have a history of allogeneic hematopoietic stem cell transplantation or organ transplantation.
* Have a history of serious Grade ≥3 immune-related adverse events (irAEs) or irAEs that led to discontinuation of a prior immunotherapy. Participants with a history of Grade ≥3 irAEs that did not lead to discontinuation of a prior immunotherapy may be included at the discretion of the investigator. If required by the investigator, after consultation with the sponsor.
* Have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently).

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence of DLTs | up to 28 days post IMP administration on Day 1 of Cycle 1 or the day before Cycle 3 Day 1, whichever comes earlier (each cycle is 14 days)
  Per dose group. During the DLT observation period.
Occurrence of treatment emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) | from first IMP administration up to 100 days after last dose of IMP or until a new anticancer therapy is initiated
  Per dose group. Assessed according to (US National Cancer Institute) Common Terminology Criteria for Adverse Events version 5.0, including Grade ≥3, serious, fatal TEAE by relationship.
Occurrence of dose interruption or discontinuation of study treatment due to TEAEs | from first IMP administration up to 14 days after the last dose of IMP
  Per dose group.
MTD or the recommended phase two dose (RP2D) of BNT317 | For MTD, up to 28 days post IMP administration on Cycle 1 Day 1 or the day before Cycle 3 Day 1, whichever comes earlier (each cycle is 14 days) or, for RP2D, up to 100 days

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | from first IMP administration up to 100 days after last dose of IMP or until a new anticancer therapy is initiated
  Per dose group. Defined as the proportion of participants in whom a complete response (CR) or partial response (PR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v1.1]) is observed as best overall response.
Duration of Response (DOR) | from first IMP administration up to 100 days after last dose of IMP or until a new anticancer therapy is initiated
  Per dose group. Defined as the time from first objective response (CR or PR per RECIST v1.1) to first occurrence of objective tumor progression (progressive disease per RECIST v1.1) or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | from at least 6 weeks after the first IMP dose up to 100 days after last dose of IMP or until a new anticancer therapy is initiated
  Per dose group. Defined as the proportion of participants with confirmed CR or PR or stable disease (per RECIST v1.1) is observed as best overall response.
PK assessment: The maximum (peak) serum concentration (Cmax) of BNT317 | from pre-dose Cycle 1 to pre-dose Cycle 4 (each cycle is 14 days)
  Per dose group. If data permits.
PK assessment: Time to reach maximum (peak) serum concentration (Tmax) of BNT317 | from pre-dose Cycle 1 to pre-dose Cycle 4 (each cycle is 14 days)
  Per dose group. If data permits.
PK assessment: Elimination half-life associated with the terminal slope of a semi-logarithmic concentration-time-curve (t1/2) of BNT317 | from pre-dose Cycle 1 to pre-dose Cycle 4 (each cycle is 14 days)
  Per dose group. If data permits.
PK assessment: The area under the curve (AUC) from time zero to infinity (mass × time × volume-1) (AUCinf) of BNT317 | from pre-dose Cycle 1 to pre-dose Cycle 4 (each cycle is 14 days)
  Per dose group. If data permits.
PK assessment: The AUC from time zero to the end of the dosing period of BNT317 | from pre-dose Cycle 1 to pre-dose Cycle 4 (each cycle is 14 days)
  Per dose group. If data permits.
The proportion of participants who are anti-drug antibody (ADA) positive against BNT317 | from first IMP administration up to 100 days after last dose of IMP or until a new anticancer therapy is initiated
  During the study.

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (11):
- United States (7):
  - Norton Cancer Institute PARENT, Louisville, Kentucky
  - START Midwest, Grand Rapids, Michigan
  - Carolina BioOncology Institute, LLC, Huntersville, North Carolina
  - Rhode Island Hospital, East Providence, Rhode Island
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Mary Crowley Cancer Research, Dallas, Texas
  - South Texas Accelerated Research Therapeutics (START), LLC, San Antonio, Texas
- Australia (4):
  - Tasman Oncology Research Ltd, Southport, Queensland
  - Cancer Research SA, Adelaide
  - Monash Medical Centre Clayton, Clayton
  - Scientia Clinical Research, Randwick

IPD SHARING:
Plan to Share IPD: No